CLINICAL TRIAL: NCT00139373
Title: Study of the Distractibility Syndrome in Patients With Progressive Supranuclear Palsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RBM0323
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2005-07

CONDITIONS: Supranuclear Palsy, Progressive
Keywords: Progressive supranuclear palsy; Frontal lobe; Oculomotor testing; Neuropsychological scores; Motor disability (UPDRS); Distractibility
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Donepezil

INTERVENTIONS:
Drug: donepezil

SUMMARY:
The syndrome of distractibility is a behavioral disorder induced by a lesion or a dysfunction of the frontal lobe. This sign is frequent in patients with progressive supranuclear palsy (PSP), a neurodegenerative disorder with severe neuronal loss in the prefrontal cortex and cholinergic systems, in particular in the Meynert basalis nucleus. This could participate in the occurrence of the distractibility in these patients. The aim of this study is to evaluate the effect of the donepezil, an anticholinesterase, on the distractibility in PSP patients, by using oculomotor and neuropsychological assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PSP
* Age > 30 years old
* Disease duration < 5 years
* Mini mental state (MMS) > 24
* Antisaccades %: 40-80%

Exclusion Criteria:

* Other parkinsonian syndromes
* MMS < 24

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Gaymard, MD, PhD, Principal Investigator — INSERM-U679
Locations (1):
- Centre d'Investigation Clinique-HÔPITAL PITIÉ-SALPETRIERE, Paris, France